CLINICAL TRIAL: NCT04447313
Title: Telephone Delivered Weight Loss, Nutrition, Exercise Study (WeLNES)
Brief Title: Telephone Delivered Weight Loss, Nutrition, Exercise WeLNES Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG1007177; NCI-2020-01624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10404 (Other: Fred Hutch/University of Washington Cancer Consortium); R01DK124114 (NIH)
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Obesity-Related Malignant Neoplasm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (ACT) (Experimental): Participants receive ACT telephone coaching over the course of 12 months, calls 1-16 weekly, calls 17-23 biweekly, and calls 24-25 monthly. Call 1 is 30 minutes in duration, while calls 2-25 are each 15-20 minutes in duration.
  Interventions: Other: Survey Administration; Behavioral: Telephone-Based Intervention
- Arm II (SBT) (Active Comparator): Participants receive SBT telephone coaching over the course of 12 months, calls 1-16 weekly, calls 17-23 biweekly, and calls 24-25 monthly. Call 1 is 30 minutes in duration, while calls 2-25 are each 15-20 minutes in duration.
  Interventions: Other: Survey Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Survey Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive ACT telephone coaching
  Arms: Arm I (ACT)
Behavioral: Telephone-Based Intervention — Receive SBT telephone coaching
  Arms: Arm II (SBT)

SUMMARY:
This phase III trial compares telephone delivered Acceptance and Commitment Therapy to standard behavioral therapy for improving weight loss in overweight or obese participants. Acceptance and Commitment Therapy focuses on increasing willingness to experience physical cravings, emotions, and thoughts while making values-guided committed behavior changes. Acceptance and Commitment Therapy may work better at improving weight loss compared to standard behavioral therapy.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive ACT telephone coaching over the course of 12 months, calls 1-16 weekly, calls 17-23 biweekly, and calls 24-25 monthly. Call 1 is 30 minutes in duration, while calls 2-25 are each 15-20 minutes in duration.

ARM II: Participants receive SBT telephone coaching over the course of 12 months, calls 1-16 weekly, calls 17-23 biweekly, and calls 24-25 monthly. Call 1 is 30 minutes in duration, while calls 2-25 are each 15-20 minutes in duration.

Participants are followed up at 6, 12, and 24 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (body mass index [BMI] >= 27) but not heavier than BMI of 45.5 (measured by weight & height)
* Wants to lose weight in the next 30 days
* Interested in learning skills to lose weight
* Willing to be randomly assigned to either condition
* Resides in United States (US)
* Has daily access to their own phone and email
* Does not have a medical or psychiatric condition that would limit their ability to comply with the behavioral recommendations of the program or pose a risk to the participant during weight loss, including meeting criteria for binge eating disorder, and meeting criteria for severe depression (CESD >= 25), or a diagnosis of serious heart disease, diabetes, uncontrolled hypertension, or cancer without written confirmation of approval from their physician office
* Not pregnant, planning to become pregnant or breastfeeding in the next 12 months
* In the past 3 months changed the dosage of prescription medications that can cause a significant change in weight or appetite
* Have not lost more than 5% of their weight in the past 6 months
* Willing and able to read in English
* Not participating in or planning to participate in other weight loss programs
* Has not participated in our other ACT intervention studies
* Does not meet criteria for combined heavy plus binge drinking
* Has access to a Bluetooth-enabled device and Wi-Fi and/or data plan
* Is not planning to have or has not recently had (past 12 months) bariatric surgery
* For outcome data retention, eligibility criteria included: Willing to complete follow-up surveys, and provide email, phone, and mailing address

Exclusion Criteria:

* The reverse of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2025-11-09 (Actual); Study Completion 2026-11-09 (Estimated)

PRIMARY OUTCOMES:
10% or more weight loss | At 12 months after randomization
  Will be measured remotely by cellular-enabled scales. Will compare the two telephone interventions, using logistic regression.

SECONDARY OUTCOMES:
Percent weight change | At 6, 12, and 24-months post randomization
  Will be measured remotely by cellular-enabled scales.
Dietary intake | At 6, 12, and 24-months post randomization
  Will be measured with the Fitbit smartphone app food logging feature.
Physical activity | At 6, 12, and 24-months post randomization
  Will be measured with the Fitbit Inspire mailed to participants.
Trajectories of weight change | At 6, 12, and 24-months post randomization
  Will compare between the two arms, with time as the independent variable using mixed effects modeling with linear, quadratic, and cubic effects of time.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Bricker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT04447313/ICF_000.pdf